CLINICAL TRIAL: NCT06994143
Title: A Phase I, Open-Label Study of CLN-978 in Patients With Treatment-Refractory Rheumatoid Arthritis (RA)
Brief Title: A Study of CLN-978, a Subcutaneously Administered CD19-directed T Cell Engager, in Subjects With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullinan Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-978-RA-101
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: RA; Treatment-refractory RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Dose Escalation (Experimental): Patients with RA treated with CLN-978 in dose escalation cohorts
  Interventions: Drug: CLN-978
- Part B Further Dose Evaluation (Experimental): Further evaluation of CLN-978 treatment of patients with RA
  Interventions: Drug: CLN-978

INTERVENTIONS:
Drug: CLN-978 — Specified dose on specified days

SUMMARY:
A Phase I, open-label study of CLN-978 in patients with treatment-refractory rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of RA which fulfills the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria ≥12 weeks prior to screening.
* Evidence of B-cell-driven disease at Screening or previous medical documentation, defined as either (i) seropositivity for RF and/or any AMPA and/or (ii) a synovial biopsy showing B-cell infiltration
* Active RA disease, as demonstrated by a DAS28 - ESR ≥3.2 and at least one swollen joint at screening.
* Inadequate response to at least 2 targeted treatments with different mechanisms. These can include tsDMARD and/or bDMARD, after failing conventional synthetic DMARD (unless contraindicated).
* Local laboratory assessments must meet the following criteria:

  * Absolute lymphocyte count (ALC) ≥0.5 x 10^9/L
  * Peripheral CD19+ B cell count ≥25 cells/μL
  * Absolute neutrophil count (ANC) ≥1.0 x 10^9/L
  * Hemoglobin (Hgb) ≥8 g/dL
  * Platelet count ≥75 x 10^9/L
  * Estimated glomerular filtration rate (eGFR) (based on the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥30 mL/min/1.73m^2
  * Total bilirubin ≤1.5 × ULN, except patients with confirmed Gilbert's Syndrome
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN
* Concurrent corticosteroids is permitted if the dose is ≤10 mg/day prednisone equivalent in the 2 weeks prior to initiation of study treatment. Hydroxychloroquine ≤400 mg/d or chloroquine ≤ 250 mg/d is allowed.

Exclusion Criteria:

* Active inflammatory disease other than RA within 12 months prior to screening or during screening that may interfere with the study assessments. Thyroiditis or secondary Sjogren's syndrome is allowed.
* Clinical evidence of any other significant unstable or uncontrolled acute or chronic disease not due to RA which, in the opinion of the Investigator could put the patient at undue risk or confound study results.
* Prior treatment with the following:

  * Cellular therapy (e.g., chimeric antigen receptor T-cell (CAR-T) or gene therapy product directed at any target.
  * Receipt of an investigational therapy within 30 days or 5 drug-elimination half-lives (whichever is longer) prior to Day 1 and during the study.
  * Received any anti-CD19 or anti-CD20 therapy such as blinatumomab, obinutuzumab, rituximab, ocrelizumab, or ofatumumab within 3 months prior to Day 1.
  * Non-biologic DMARD within 14 days prior to Day 1.
  * Cyclophosphamide or a biologic immunomodulating therapy within 2 months of Day 1.
* Live or live-attenuated vaccines within the 4 weeks prior to the Screening visit or during the Screening Period
* Active or latent tuberculosis (TB) evidenced by a positive or indeterminant Interferon Gamma Release Assay (IGRA), unless the patient has documented previous completion of TB treatment and no current clinical indication of TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 48 wks
  Incidence and severity of adverse events (AEs)/adverse events of special interest (AESIs)/serious adverse events (SAEs)

SECONDARY OUTCOMES:
Serum concentrations of CLN-978 | 12 wks
  Serum concentrations of CLN-978
Level of anti-drug antibodies | 12 wks
  Level of anti-drug antibodies
Pharmacodynamics-related biomarker | 48 wks
  Levels of total B lymphocytes in the peripheral blood

CONTACTS AND LOCATIONS:
Locations (2):
- Cullinan Investigative Site, Erlangen, Germany
- Cullinan Investigative Site, Rome, Italy